CLINICAL TRIAL: NCT02587065
Title: Multicenter Interventional Phase IV Study for the Assessment of the Effects on Patient's Satisfaction of Plegridy (Pre-filled Pen) in Subjects With Relapsing-remitting Multiple Sclerosis Unsatisfied With Other Injectable Subcutaneous Interferons (PLATINUM)
Brief Title: Plegridy Satisfaction Study in Participants
Acronym: PLATINUM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITA-PEG-14-10779; 2015-002201-11 (EudraCT Number)
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Relapsing-Remitting Multiple Sclerosis (RRMS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — peginterferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- peginterferon beta-1a (Experimental): 125 μg administered subcutaneously (SC) every 2 weeks
  Interventions: Drug: peginterferon beta-1a

INTERVENTIONS:
Drug: peginterferon beta-1a — 125 mcg administered subcutaneously (SC) every 2 weeks.
  Other Names: BIIB017; PEGylated Interferon Beta-1a; Plegridy; PEG IFN β-1a

SUMMARY:
The primary objective of this study is to investigate whether Peg-IFN beta-1a improves the satisfaction of Relapsing-Remitting Multiple Sclerosis (RRMS) participants unsatisfied with injectable subcutaneous Interferons, as measured by the Abbreviated Treatment Satisfaction Questionnaire to Medication (TSQM-9), at 12 weeks. The secondary objectives of this study are to evaluate in this study population: effects of Peg-IFN beta-1a treatment on participants' satisfaction at 24 weeks; effects of Peg-IFN beta-1a treatment on short-term participants' adherence; effects of Peg-IFN beta-1a treatment on participants' fatigue; effects of Peg-IFN beta-1a on disease activity and physical disability; impact of Peg-IFN beta-1a treatment on participant-reported health-related quality of life; impact of Peg-IFN beta-1a treatment on participants' injection-system satisfaction; Evaluate the relationship between participants' satisfaction and adherence; Evaluate the relationship between participants' satisfaction and social-demographic factors (age, sex, employment working, level of education, etc) and clinical characteristics (annualized relapse rate [ARR], disability, etc.) and to evaluate the treatment safety and tolerability.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects diagnosed with Relapsing Remitting MS according to 2010 McDonald criteria.
* Subjects with EDSS score between 0.0 and 5.0 at baseline.

Key Exclusion Criteria:

* Pregnancy or breast-feeding.
* Have any contra-indications to treatment with Peg-IFN-beta 1a according to the Summary of Product Characteristics.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (26):
- Italy (26):
  - Research Site, Arezzo
  - Research Site, Bari
  - Research Site, Cagliari
  - Research Site, Cefalù
  - Research Site, Chieti
  - Research Site, Como
  - Research Site, Fidenza
  - Research Site, Foligno
  - Research Site, Gallarate
  - Research Site, Genova
  - Research Site, L’Aquila
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Mondovì
  - research Site, Napoli
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Ozieri
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Pietra Ligure
  - Research Site, Pozzilli
  - Research Site, Reggio Calabria
  - Research Site, Roma
  - Research Site, Torino

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 32 sites in Italy.
Pre-assignment Details: A total of 193 participants with relapsing remitting multiple sclerosis (RRMS) were enrolled into the study.
Groups:
- Peg-interferon Beta-1a 125 μg: Participants received peg-interferon beta-1a 63 μg on Day 1 followed by peg-interferon beta-1a 94 μg on Day 14 in the titration phase. Participants received per-interferon beta-1a on Day 28 and then every 2 weeks for up to 12 months.
Period: Overall Study
Arm/Group | Peg-interferon Beta-1a 125 μg
Started | 193
Completed | 166
Not Completed | 27
Not completed — Adverse Event | 14
Not completed — Withdrawal of Informed Consent (IC) | 5
Not completed — Non-adherence to the Protocol | 3
Not completed — Discontinuation of Study Medication | 2
Not completed — Reason not Specified | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population included all enrolled participants who took at least one dose of the study medication.
Arm/Group | Peg-interferon Beta-1a 125 μg
Number analyzed (Participants) | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 193
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135
  Male | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 192
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Convenience Satisfaction Score of Treatment Satisfaction Questionnaire to Medication (TSQM-9) at Week 12
Description: TSQM is a 14-item instrument consisting of four scales: effectiveness scale (questions 1 to 3), side effects scale (questions 4 to 8), convenience scale (questions 9 to 11) and global satisfaction scale (questions 12 to 14). In TSQM-9, the five items related to side effects of medication were not included. The scores were computed by adding items for each domain. The lowest possible score was subtracted from this composite score and divided by the greatest possible score minus the lowest possible score. This provided a transformed score between 0 and 1 that was then multiplied by 100. TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain. Questionnaires were completed electronically by participants, by means of a participant i-PAD at each study visit.
Time Frame: Baseline, Week 12
Population: FAS population included all enrolled participants who took at least one dose of the study medication. Number analyzed are the participants who were evaluated at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peg-interferon Beta-1a 125 μg
Number analyzed (Participants) | 193
score on a scale
  Baseline: number analyzed (Participants) | 192
  Baseline | 38.5 (13.9)
  Change at Week 12: number analyzed (Participants) | 188
  Change at Week 12 | 38.5 (23.3)
Statistical Analysis 1: Comparison: Peg-interferon Beta-1a 125 μg; Adjusted change of convenience satisfaction domain of TSQM-9; Test type: Other; p = 0.56, Mixed-effects REML regression; Spearman's correlation coefficient = -0.85, 95% CI 2-sided [-3.72 to 2.02]

2. Secondary Outcome: Change From Baseline in the Score of All Domains of TSQM-9 at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peg-interferon Beta-1a 125 μg
Number analyzed (Participants) | 193
score on a scale
  Baseline: Convenience Satisfaction: number analyzed (Participants) | 176
  Baseline: Convenience Satisfaction | 38.5 (13.9)
  Change at Week 24: Convenience Satisfaction: number analyzed (Participants) | 176
  Change at Week 24: Convenience Satisfaction | 41.9 (22.5)
  Baseline: Effectiveness: number analyzed (Participants) | 176
  Baseline: Effectiveness | 47.0 (17.5)
  Change at Week 24: Effectiveness | 21.2 (26.9)
  Baseline: Global satisfaction | 41.4 (17.3)
  Change at Week 24: Global satisfaction | 27.9 (26.1)

3. Secondary Outcome: Change From Baseline in Number of Participants With Adherence to Study Treatment at Weeks 12 and 24
Description: Adherence to treatment was evaluated using a questionnaire assessing adherence and the reasons for not taking drug at the recommended frequency of administration. Participants who had taken the prescribed doses of treatment in the previous 28 days were evaluated.
Time Frame: Baseline, Weeks 12 and 24
Population: FAS population included all enrolled participants who took at least one dose of the study medication. Overall number of participants analyzed are the participants who were evaluated for the outcome measure.
Measure: Number; unit: participants
Arm/Group | Peg-interferon Beta-1a 125 μg
Number analyzed (Participants) | 113
participants
  Baseline | 113
  Change at Week 12 | 65
  Change at Week 24 | 53

4. Secondary Outcome: Change From Baseline in Fatigue Status Scale (FSS) Score at Weeks 12 and 24
Description: FSS is a questionnaire composed of nine statements on the state of fatigue experienced during the previous week. The answers are within a scale of agreement ranging from 1 to 7, where 1 represents less fatigue and 7 indicates highest fatigue. The total score was obtained summing the number given at each item and it ranges from 7 to 63. An overall score of ≥36 indicates a state of fatigue. Questionnaires were completed electronically by participants, by means of a participant i-PAD at each study visit. Here, negative values indicate improvement in FSS score from baseline.
Time Frame: Baseline, Weeks 12 and 24
Population: FAS population included all enrolled participants who took at least one dose of the study medication. Number analyzed are the participants who were evaluated at each time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peg-interferon Beta-1a 125 μg
Number analyzed (Participants) | 193
score on a scale
  Baseline | 40.1 (15.6)
  Change at Week 12: number analyzed (Participants) | 191
  Change at Week 12 | -4.6 (13.1)
  Change at Week 24: number analyzed (Participants) | 176
  Change at Week 24 | -3.8 (13.1)

5. Secondary Outcome: Change From Baseline in Adapted Sclerosis Treatment Concerns Questionnaire (MSTCQ) Score at Weeks 12 and 24
Description: MSTCQ is a 20-item questionnaire adapted for 'Peg-interferon Beta 1a' containing two domains: injection system satisfaction (1-9) and side effects (1-11). All questions in the MSTCQ have a five-point response choice, with a minimum possible total score of 20 and a maximum possible total score of 100. Lower total scores indicating better outcomes. Questionnaires were completed electronically by participants, by means of a participant I-PAD at each study visit. Here, negative values indicate improvement in MSTCQ score from baseline.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peg-interferon Beta-1a 125 μg
Number analyzed (Participants) | 193
score on a scale
  Baseline | 71.9 (14.0)
  Change at Week 12: number analyzed (Participants) | 191
  Change at Week 12 | -16.8 (16.9)
  Change at Week 24: number analyzed (Participants) | 176
  Change at Week 24 | -19.4 (17.1)

6. Secondary Outcome: Change From Baseline in Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) Score at Week 12 and 24
Description: MusiQoL is a self-administered questionnaire consisting of 31 items describing nine dimensions of health-related quality of life (QoL): activities of daily living, psychological wellbeing, symptoms, relationship with friends, relationship with family, sentimental and sexual life, coping rejection, relationship with healthcare system). All items are scored based on frequency/extent of an event on a five-point scale ranging from never/not at all (option 1) to always/very much (option 5). Total score is obtained by linearly transforming and standardizing on a 0-100 scale. Higher scores indicate a better level of health-related QoL for each dimension and for the global index score. Here, negative values indicate improvement in MusiQoL score from baseline.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peg-interferon Beta-1a 125 μg
Number analyzed (Participants) | 193
score on a scale
  Baseline | 67.8 (16.5)
  Change at Week 12: number analyzed (Participants) | 191
  Change at Week 12 | 4.6 (14.89)
  Change at Week 24: number analyzed (Participants) | 176
  Change at Week 24 | 5.0 (14.2)

7. Secondary Outcome: Change From Baseline in Annualized Relapse Rate (ARR) at Week 24
Description: Relapses are defined as neurologic symptoms lasting more than 24 hours which occur at least 30 days after the onset of a preceding event. ARR was calculated as the total number of relapses for all participants divided by the total participant-years of exposure to that treatment. Here negative sign indicates decrease in annual relapse rate as compared to baseline.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Number; unit: relapses per participant-year
Arm/Group | Peg-interferon Beta-1a 125 μg
Number analyzed (Participants) | 193
relapses per participant-year
  Baseline | 0.15
  Change at Week 24: number analyzed (Participants) | 176
  Change at Week 24 | -0.03

8. Secondary Outcome: Percent Change in Relapse-Free Participants at Week 24
Description: Relapses are defined as neurologic symptoms lasting more than 24 hours which occur at least 30 days after the onset of a preceding event. Percent change in relapse-free participants had been calculated with respect to the number of relapse-free participants at baseline. Here, negative sign indicates decrease in number of relapse free participants at specified timepoint as compared to baseline.
Time Frame: Baseline, Week 24
Population: FAS population included all enrolled participants who took at least one dose of the study medication. Number of participants analyzed are the participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage change
Arm/Group | Peg-interferon Beta-1a 125 μg
Number analyzed (Participants) | 189
percentage change | -7.94

9. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can herefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Baseline up to Week 24
Population: FAS population included all enrolled participants who took at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Peg-interferon Beta-1a 125 μg
Number analyzed (Participants) | 193
Participants | 82

10. Secondary Outcome: Number of Participants With AE Stratified by Severity
Description: Severity of AEs was evaluated based on the following criteria- Mild: Symptoms barely noticeable to participant or does not make participant uncomfortable; does not influence performance or functioning; prescription drug not ordinarily needed for relief of symptom(s) but may be given because of personality of participant. Moderate: Symptoms of a sufficient severity to make participant uncomfortable; performance of daily activity is influenced; participant is able to continue in study; treatment for symptom(s) may be needed. Severe: Symptoms cause severe discomfort; symptoms cause incapacitation or significant impact on participant's daily life; severity may cause cessation of treatment with study treatment; treatment for symptom(s) may be given and/or participant hospitalized.
Time Frame: Baseline up to Week 24
Population: FAS population included all enrolled participants who took at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Peg-interferon Beta-1a 125 μg
Number analyzed (Participants) | 193
Participants
  Mild | 55
  Moderate | 27

11. Secondary Outcome: Number of Participants With Clinical Abnormal Laboratory Values
Description: Participants with clinical abnormal laboratory values were reported throughout the studies.
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Peg-interferon Beta-1a 125 μg
Number analyzed (Participants) | 193
Participants
  Baseline | 4
  Week 12: number analyzed (Participants) | 191
  Week 12 | 3
  Week 24: number analyzed (Participants) | 176
  Week 24 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Description: FAS population included all enrolled participants who took at least one dose of the study medication.
Arm/Group | Peg-interferon Beta-1a 125 μg
All-Cause Mortality (participants affected / at risk) | 0/193
Serious Adverse Events (participants affected / at risk) | 0/193
Other Adverse Events (participants affected / at risk) | 44/193
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peg-interferon Beta-1a 125 μg (N=193)
Influenza like illness (General disorders) | 28 (42)
Injection site reactions (General disorders) | 10 (12)
Pyrexia (General disorders) | 10 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2015-07-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT02587065/Prot_001.pdf
  • Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT02587065/SAP_000.pdf